CLINICAL TRIAL: NCT00226083
Title: Studies of Large Platelets in Patients With Sickle Cell Disease
Brief Title: Study of Blood Platelets in Sickle Cell Disease
Status: Withdrawn | Type: Observational
Why Stopped: PI returned to India
Sponsor: Rockefeller University (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other); Schneider Children's Hospital of North Shore (Other)
Responsible Party: Sponsor
Other Study IDs: RUH IRB # AST-0565-0805
Record Dates: First submitted 2005-09-22; First posted 2005-09-26 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
We are studying if sickle cell disease blood platelets are larger than normal and how they may cause obstruction of blood vessels. We are also trying to study the reasons why large platelets are found in patients with sickle cell disease.

DETAILED DESCRIPTION:
Research volunteers are seen in the Outpatient Research Center by the Principal Investigator or another physician. A detailed history is obtained, a physical examination is performed, and blood (usually 4 tablespoons) is obtained for additional tests. The research volunteer's previous medical records will be requested. Upto 5 additional blood samples may be obtained in a subgroup of patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults and children > 7 years of age with sickle cell disease (Hb SS) who are not taking hydroxyurea and are not receiving routine blood transfusion therapy.

Exclusion Criteria:

* Current hydroxyurea therapy or,
* Hydroxyurea use within the past 3 months
* Blood transfusion or exchange transfusion within the past 3 months
* Current treatment with aspirin or clopidogrel

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adults and children with sickle cell disease (Hb SS)
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2005-08; Primary Completion 2007-09 (Estimated); Study Completion 2007-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Arun Shet, MD, Principal Investigator — Rockefeller University
Locations (1):
- Rockefeller University Hospital, New York, New York, United States